CLINICAL TRIAL: NCT00370123
Title: In This Study we Aim to Explore the Immune Nature of Endometriosis as Manifested in the Peripheral Blood, Endometriosis Lesions, Normal Peritoneum and Normal Endometrium of Patients Suffering From Documented Endometriosis.
Brief Title: The Immune Base of Endometriosis
Status: Withdrawn | Type: Observational
Why Stopped: The study was withrawn do to logistic difficulties
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4251-RM-CTIL
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Endometriosis
Keywords: endometriosis; apoptosis; regulatory T cells
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Endometriosis is a chronic disabling inflammatory disease which effects 15-20% of women in their reproductive life.

In patients suffering from endometriosis retrograded menstrual cells induce an inflammatory response.Endometriosis has also been considered to be an autoimmune disease, owing to the presence of auto antibodies, the association with other autoimmune diseases and recurrent immune-mediated abortion.

We aim to study this aberrant regulation of endometrial cell apoptosis by investigating the peripheral blood immune system of patients suffering from endometriosis.

Hypothesis:

We hypothesized that immune peripheral mononuclear cells of patients suffering from pelvic endometriosis react differently to eutopic endometrial cells than matched control women group. This difference could be study on a molecular, antigenic and/or apoptotic cycle gene expression. We also hypothesized that a deficiency of regulatory T cells is associated with the progression of endometriosis.

DETAILED DESCRIPTION:
Endometriosis affects 15-20% of women in their reproductive life. Endometriosis is a chronic disabling inflammatory disease, characterized by implantation and growth of endometrial tissue (glandular epithelium and stroma) outside the uterine cavity.

Retrograde menstruation was found in 80%-90% of women. In most women these endometrial cells undergo apoptosis. In patients suffering from endometriosis this cells induce an inflammatory response. Pelvic endometriosis is associated with intrinsic anomalies of the refluxed endometrium, increased secretion of pro-inflammatory cytokines, neoangiogenesis, and impaired function of cell-mediated natural immunity.

Endometriosis has also been considered to be an autoimmune disease, owing to the presence of auto antibodies, the association with other autoimmune diseases and recurrent immune-mediated abortion.

Evidence suggests that Foxp3-expressing CD4+CD25+ regulatory T cells play a crucial role in the suppression of inflammatory disease. However, their role in the suppression of endometriosis has not yet been addressed.

We aim to study this aberrant regulation of endometrial cell apoptosis by investigating the peripheral blood immune system of patients suffering from endometriosis.

Hypothesis:

We hypothesized that immune peripheral mononuclear cells of patients suffering from pelvic endometriosis react differently to eutopic endometrial cells than matched control women group. This difference could be study on a molecular, antigenic and/or apoptotic cycle gene expression. We also hypothesized that a deficiency of regulatory T cells is associated with the progression of endometriosis.

Study design:

This is an open labeled prospective in vitro study for two years.

Patients:

50 Patients suffering from endometriosis undergoing laparoscopy will be compared to 50 patients undergoing laparoscopy for other reasons.

Methods:

1. Blood withdrawal and pipelle endometrial cells harvesting 2. Isolation of peripheral blood mononuclear cells (PBMC) 3. Generation of T cell lines (from patients) 4. Measurement of cytokines 5. Determination of T- cell subsets by flow cytometry 5. PMNC and T cell lines will be frozen in liquid nitrogen and stored at-70C for future studies.

6. Endometrial tissue will be served ad antigenic source to generated T cell lines and the remnants will be stored at-70C for future studies.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopically proven endometriosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women of childbrearing age suffering from endometriosis and undergoing laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Mati Mandel, MD, Study Chair — Sheba Medical Center